CLINICAL TRIAL: NCT01240213
Title: Vitamin D, Weight Loss, and Breast Cancer Biomarkers
Brief Title: Vitamin D, Diet and Activity Study
Acronym: ViDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Anne McTiernan, MD PhD, FHCRC
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SAC110024; IR 7297 (Other: FHCRC IRB)
Record Dates: First submitted 2010-11-09; First posted 2010-11-15 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer; Obesity; Hypovitaminosis D
Keywords: Vitamin D; lifestyle intervention; postmenopausal women
MeSH Terms: conditions — Breast Neoplasms; Obesity; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): 2000 IU per day of Vitamin D
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 2000 IU per day of Vitamin D
  Other Names: calciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — 1 Placebo per day
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Experimental and human data suggests that vitamin D could protect against breast cancer. Overweight/obese individuals are at increased risk of low vitamin D levels. Vitamin D may reduce production of fat tissue, thereby reducing weight gain, which would result in lower levels of adipose-derived hormones and other breast cancer risk factors.The purpose of this study is to test the effect of vitamin D supplementation on the response to a weight loss (diet + exercise) intervention and select breast cancer risk factors in overweight and obese postmenopausal women with low blood vitamin D levels.

DETAILED DESCRIPTION:
Objective: To test the incremental effect of vitamin D supplementation (2000 IU/day) in 228 overweight and obese postmenopausal women with low blood vitamin D levels on response to a weight loss (diet + exercise) intervention in a double-blind placebo-controlled clinical trial.

Primary Aim:

• Determine the effects of 12-months vitamin D supplementation vs. placebo on weight loss in women following a weight loss diet and exercise program.

Secondary Aims:

* Determine the effects of 12-months vitamin D vs. placebo on blood biomarkers associated with increased breast cancer risk (insulin, glucose, CRP).
* Test 12-months vitamin D effects on muscle strength as measured by 1RM leg press and bench press in women undergoing weight loss.
* Test the effect of 12-month vitamin D supplementation on effects on quality of life (QOL) in women undergoing weight loss.

Additional Aims:

* In a 50% subset of women, test the effect of 12-month vitamin D supplementation vs. placebo on breast epithelial cell cytomorphology (quantified by the Masood cytology index) obtained through random periareolar fine needle aspiration (RPFNA).
* Collect subcutaneous abdominal fat aspirations in the 50% subsample of women.

OUTLINE: This is a randomized study. Participants are stratified according to body mass index (< 30 vs ≥ 30) and RPFNA-consent. All participants will receive a 6-month weight loss intervention (prescribed weight loss goal of 10% of initial body weight) followed by 6 months' maintenance therapy.

Baseline, 6-, and 12-month measurements will include weight, BMI, waist and hip circumference, serum 25-hydroxyvitamin D, fasting blood samples, and questionnaires on details of diet especially items containing vitamin D, physical activity levels, sun exposure including clothing and sunscreen habits, dietary supplement and vitamin use, and medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years
* Postmenopausal (no periods for past 12 months)
* Screening serum vitamin D (25(OH)D) between 10 and 32 ng/mL ("insufficient")
* No menopausal HRT use of any type including vaginal X 6 months and willing to avoid use for study duration
* BMI > 25.0 kg/m2 (> 23.0 for Asians)
* Physically able to undertake a calorie reduction and exercise program
* Able to come for clinic visits, classes, and measurements, fill out questionnaires and logs in English
* Gives informed consent, agrees to be randomly assigned

Exclusion Criteria:

* Currently using more that 400 IU vitamin D from supplemental sources
* Screening vitamin D level < 10 ng/mL (will be referred to primary provider) or > 32 ng/mL (already sufficient)
* Osteoporosis
* Renal disease, history of kidney stones
* Any contra-indications to taking vitamin D 2000 IU/day
* Plans to leave the study area within the follow-up period
* Plans to join another organized weight loss program or take appetite suppressant medication during the study period
* History of bariatric surgery
* Current use of medications likely to interfere with adherence to interventions or study outcomes
* Current smoker
* Personal history of invasive or in situ breast cancer
* Personal history of invasive cancer other than breast: except for non- melanoma skin cancer which would be eligible
* Diabetes mellitus
* Abnormalities on screening physical that contraindicate participation
* Severe congestive heart failure per NYHA criteria 3 & 4
* Contraindications for entry into a research exercise program: recent (within 6 months) myocardial infarction, pulmonary edema, myocarditis, pericarditis, unstable angina, pulmonary embolism, deep vein thrombosis, uncontrolled hypertension (systolic > 200, diastolic > 100), orthostatic hypotension, moderate/severe aortic stenosis, uncontrolled arrythmia, uncontrolled congestive heart failure, left bundle branch block, history of cardiac arrest or stroke
* Alcohol or drug abuse, significant mental illness (as assessed by study staff impression)
* For the RPFNA/adipose tissue substudy: bilateral breast cancer, bilateral mastectomy, unable or unwilling to stop aspirin or NSAIDs for 1 week before and after the procedure, allergy to anesthetics or local anesthetics.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Compare the effects of a 1-year one year Vitamin D supplementation vs placebo, on weight loss in postmenopausal women following a weight loss diet and exercise program. | One Year

SECONDARY OUTCOMES:
Determine the effects of 12-months vitamin D vs. placebo on blood biomarkers (insulin,glucose,CRP) associated with increased breast cancer risk. | One Year
Test 12-months vitamin D effects on muscle strength as measured by 1RM leg press and bench press in women undergoing weight loss. | One Year
Test the effect of 12-month vitamin D supplementation on effects on quality of life (QOL) in women undergoing weight loss. | One Year
Effect of Vitamin D supplementation on breast epithelial cell cytomorphology | One Year
  In a 50% subset of women, test the effect of 12-month vitamin D supplementation vs. placebo on breast epithelial cell cytomorphology (quantified by the Masood cytology index) obtained through random periareolar fine needle aspiration (RPFNA).
Effect of Vitamin D on epithelial cell gene expression | One year
  In a 50% subset of women, test the effect of 12-month vitamin D supplementation vs. placebo on breast epithelial cell gene expression as measured by qRT-PCR. The breast epithelial cells are collected by RPFNA

CONTACTS AND LOCATIONS:
Overall Officials: Anne McTiernan, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Mason C, de Dieu Tapsoba J, Duggan C, Wang CY, Korde L, McTiernan A. Repletion of vitamin D associated with deterioration of sleep quality among postmenopausal women. Prev Med. 2016 Dec;93:166-170. doi: 10.1016/j.ypmed.2016.09.035. Epub 2016 Sep 28. PMID 27687537
- [Derived] Mason C, Tapsoba JD, Duggan C, Imayama I, Wang CY, Korde L, McTiernan A. Effects of Vitamin D3 Supplementation on Lean Mass, Muscle Strength, and Bone Mineral Density During Weight Loss: A Double-Blind Randomized Controlled Trial. J Am Geriatr Soc. 2016 Apr;64(4):769-78. doi: 10.1111/jgs.14049. Epub 2016 Apr 5. PMID 27060050
- [Derived] Duggan C, de Dieu Tapsoba J, Mason C, Imayama I, Korde L, Wang CY, McTiernan A. Effect of Vitamin D3 Supplementation in Combination with Weight Loss on Inflammatory Biomarkers in Postmenopausal Women: A Randomized Controlled Trial. Cancer Prev Res (Phila). 2015 Jul;8(7):628-35. doi: 10.1158/1940-6207.CAPR-14-0449. Epub 2015 Apr 23. PMID 25908506
- [Derived] Mason C, Xiao L, Imayama I, Duggan C, Wang CY, Korde L, McTiernan A. Vitamin D3 supplementation during weight loss: a double-blind randomized controlled trial. Am J Clin Nutr. 2014 May;99(5):1015-25. doi: 10.3945/ajcn.113.073734. Epub 2014 Mar 12. PMID 24622804